CLINICAL TRIAL: NCT02689908
Title: Individualized Radiation Dose Control: Could Neck Circumference be a New Somatometric Parameter to Adjust Tube Current for Thorax CT?
Brief Title: Individualized Radiation Dose Control
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Van Military Hospital (Other Government)
Responsible Party: Principal Investigator, ferhat, staff radiology specialist, department of radiology, Van Military Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: VETH123
Record Dates: First submitted 2016-01-31; First posted 2016-02-24 (Estimated); Last update posted 2016-02-24 (Estimated); Status verified 2016-02

CONDITIONS: Radiation Exposure
Keywords: Thorax CT; Low Dose; Body Mass Index; Neck Circumference

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- The patients underwent thorax CT (Other): The patients refered to radiology service underwent thorax computed tomography without contrast material for the evaluation of various complaints such as dyspnea, hemoptysis and pulmonary infections.
  Interventions: Radiation: computed tomography

INTERVENTIONS:
Radiation: computed tomography — low dose protocol of thorax ct

SUMMARY:
The adjustment of radiation dose in many CT protocol are based on body mass index(BMI) or weight of the patient.

In the literature, neck circumference (NC) has been reported as a new anthropometric parameter indicating the body mass for the upper body.

NC may be an important landmark in the determination of the low dose protocols for upper body CT examinations such as neck, chest and coronary CT.

DETAILED DESCRIPTION:
Over the last few decades, MDCT(multidetector computed tomography), cardiac imaging, CT perfusion techniques, high-pitch CT, and dual-energy CT have been introduced to clinical practice, increasing the overall amount of radiation applied. There are two types of approaches in accordance with the "as low as reasonably achievable (ALARA)" principle in MDCT. One of them is related to new technology products and different imaging techniques such as dose modulation along the x-, y-, and z-axes (anatomical tube current modulation, ECG-controlled tube current modulation or dynamically adjustable pre-patient collimation of the X-ray beam in the z-axis direction, iterative reconstruction technique. The other strategy is individualized screening-dose protocols based on body size. However the radiologist is facing the challenge of providing diagnostic image quality at the lowest radiation dose.

Body mass index (BMI) is not only the most widely used anthropometric tool for defining overweight and obesity, but it is also the most commonly reported body index for adjusting low dose in MDCT.Despite this popularity of BMI, it is becoming increasingly more clear that BMI is not a good surrogate for regional adiposity. Regional fat deposition, especially in the upper body region, is a better predictor of some obesity related complications than BMI. Accordingly, it has been reported that several anthropometric parameters of the chest might serve as a surrogate instead of BMI for individualized dose settings Neck circumference(NC) is a kind of somatometric parameter like wrist or hip circumference that reflects the upper body size. NC may be an important landmark in the determination of the low dose protocols for upper body CT examinations such as neck, chest and coronary CT. Although investigators have not encountered studies in the literature, this point will be evaluated in our study.The purpose of this study is to evaluate if NC is an appropriate and a novel parameter for adjusting and reduction of the effective chest CT radiation doses in comparison with BMI or not.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of pulmonary diseases
* participants who can be referred to radiology for diagnostic imaging
* participants who allowed to be taken somatometric measurements

Exclusion Criteria:

* participants who did not allow to be taken somatometric measurements
* participants with incomplete data (such as missing weight or height data)
* pediatric and pregnant patients

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-05; Primary Completion 2016-02 (Estimated); Study Completion 2016-02 (Estimated)

PRIMARY OUTCOMES:
The measurement of neck circumference of the patients undergoing non-enhanced thorax CT | 1 year
  Before CT examination, during patient preparation, neck circumference was measured horizontally at the level of the cyricoid cartilage by a non-elastic flexible tape (centimeter, cm)

SECONDARY OUTCOMES:
The measurement of weight of the patients undergoing non-enhanced thorax CT | 1 year
  Before CT examination, during patient preparation, patient weight was measured by a bascule (kilogram, kg)
The measurement of height of the patients undergoing non-enhanced thorax CT | 1 year
  Before CT examination, during patient preparation, patient height was measured with a stadiometer (milimeter, mm)
Calculating the body mass index (BMI) using the results of each patient measured in outcome 2 and outcome 3. | 1 year
  calculation of data with a spesific formula (kg/mm²)

CONTACTS AND LOCATIONS:
Overall Officials: serkan arıbal, Principal Investigator — Aksaz Military Hospital
Locations (2):
- Turkey (Türkiye) (2):
  - Ferhat, Van, Van
  - Erdem, Van, Van

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Ghoshhajra BB, Engel LC, Major GP, Verdini D, Sidhu M, Karolyi M, Abbara S, Hoffmann U, Kalra M, Brady TJ. Direct chest area measurement: A potential anthropometric replacement for BMI to inform cardiac CT dose parameters? J Cardiovasc Comput Tomogr. 2011 Jul-Aug;5(4):240-6. doi: 10.1016/j.jcct.2011.06.003. Epub 2011 Jun 12. PMID 21723515
- See also: a similar study in the literature — http://www.ncbi.nlm.nih.gov/pubmed/21723515